CLINICAL TRIAL: NCT05090943
Title: Adult Tic Disorders Registry
Acronym: RegisTICs
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210801
Record Dates: First submitted 2021-09-22; First posted 2021-10-25 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Tic Disorders
MeSH Terms: conditions — Tic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Quality of life questionnaires
  Interventions: Other: QOL to be completed by the participant

INTERVENTIONS:
Other: QOL to be completed by the participant — The scales (PUTS, OCI, TS-QOL, ASRS, GAD-7, PHQ9, TAPS) to be completed by the participant

SUMMARY:
The purpose of this study is to develop the adult tic disorders registry in order to characterize the relationship between tic severity and tic-related impairment in women compared to men with tic disorders.

ELIGIBILITY:
Inclusion criteria :

1. Age >18 years
2. Patients with Tic disorders
3. Given the non-opposition

Non Inclusion criteria

1. No affiliation to a French health social insurance
2. Significant congenital disorders that may affect understanding of assessments
3. Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with tics disorders
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between Quality of Life and TICs severity | 6 months
  Severity of the tics measurement (YGTSS Impairment Score) and the quality of life (TS-QOL) between men and women with tic disorders, while controlling for the YGTSS Total Tic Score

SECONDARY OUTCOMES:
Change in TICs | 6 months
  Change in tic inventories/tic migrations with the YGTSS tic inventories

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Limoges, Limoges
  - CHU Marseille, Marseille
  - Service de Neurologie, GH Pitié Salpêtrière, Paris
  - CHU Poitiers, Poitiers
  - CHU Nantes, Saint-Herblain
  - CHU Strasbourg, Strasbourg